CLINICAL TRIAL: NCT02904941
Title: Human Amniotic Versus Synthetic Membrane as a Transient Skin Cover for Pediatric Burns: A Randomised Trial
Brief Title: Human Amniotic Versus Synthetic Membrane as a Transient Skin Cover for Pediatric Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other); Hospital Carlos Van Buren (Other)
Responsible Party: Principal Investigator, Sandra Montedonico Rimassa, MD, PhD, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA15I20099
Record Dates: First submitted 2016-09-04; First posted 2016-09-19 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Burns
Keywords: Children; Skin Transplantation; Amniotic Membrane
MeSH Terms: conditions — Burns | interventions — Biological Dressings

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amniotic Membrane Dressing (Experimental): Children allocated to this arm will receive skin dressings made out of human amniotic membrane. Dressings will be replaced every 72 - 96 hours.
  Interventions: Biological: Amniotic Membrane Dressing; Procedure: Standard Wound Care
- Synthetic Dressing (Active Comparator): Children allocated to this arm will receive skin dressings made out of silicone as part of their wound care. Dressings will be replaced every 72 - 96 hours.
  Interventions: Device: Synthetic Dressing; Procedure: Standard Wound Care

INTERVENTIONS:
Biological: Amniotic Membrane Dressing — Amniotic membrane dressings will be made out of donated amniotic membranes from elective cesarean sections. Screening for relevant infectious diseases and irradiation will be performed from every included sample in order to minimise infectious risks. Dressings will be provided to attending surgeons during wound care at the operating theatre and removed every 72-96 hours.
  Arms: Amniotic Membrane Dressing
Device: Synthetic Dressing — Silicone dressings will used as an active comparator in this study. As with the amniotic membrane, dressings will be applied to wound care at the operating room and replaced every 72 to 96 hours.
  Other Names: Mepitel (R)
  Arms: Synthetic Dressing
Procedure: Standard Wound Care — Every included participant will receive standard wound care regardless of treatment allocation. Contaminants such as clothes or other materials will be removed, and all burns will be cleaned using sterile saline solutions. Clorhexidine will also be used to clean the skin. Surgical debridement under general anesthesia or procedural sedation/analgesia will be performed to every included participant, in which nonviable tissues and blisters will be removed.

SUMMARY:
This is a randomised trial that aims to evaluate whether a transient skin cover made out of human amniotic membranes is effective in managing burns among pediatric patients. The primary outcome of this trial is the proportion of skin grafted amongst participants. Secondary outcomes include hospital stay and the number of surgical debridements required by included patients.

DETAILED DESCRIPTION:
Patients with burns that compromise 5% or more of total body surface area will be randomised to receive a membrane made out of human amnios or a synthetic cover for the acute phase of care. Eligible participants will be children with acute burns (<24 hours) due to hot liquids that compromise 5% or more of total body surface area.

Patients with burns due to fire, hot surfaces or chemical agents, those with delayed presentation to the emergency department (>24 hours), and patients with burns that compromise the head or scalp (exclusively or in cases where this compromise exceeds 50% of the total body surface area affected by the burn). Patients whose parents do not authorise participation in this trial will also be excluded.

Randomisation will be performed by a statistician unaware of the clinical management of included patients. The specific allocation sequence will be kept hidden from other investigators. Patients, outcome assessors and statisticians will also be kept unaware of treatment allocation. Blinding will be achieved by using image analysis software to assess the primary endpoint. Due to the intervention's characteristics, it will be impossible to perform blinding of the attending surgeon. Analyses will be performed under the intention - to - treat principle.

Amniotic membrane samples will be collected by personnel that shall not provide care for included participants. Samples suitable for donation will come from elective caesarean sections. Once obtained, amniotic membranes will be stored in sterile containers and then sent for irradiation at a facility provided by the Comisión Chilena de Energía Nuclear (Chilean Nuclear Energy Comission). This sampling protocol includes exclusion of relevant infectious diseases as established by the Chilean Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Children with an acute burn (<24 hours)
* Burn due to hot liquids.
* Total wound extension at least 5% of total body surface area.

Exclusion Criteria:

* Burns due to fire, chemical burns or hot surfaces.
* Delayed burns (>24 hours).
* Burns extending solely to the head or scalp.
* Burns whose compromise of head or scalp is 50% or more of total burn area.
* Refusal to participate.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total Grafted Skin Area | Within the first 30 days after randomisation

SECONDARY OUTCOMES:
Length of Hospital Stay | Within the first 45 days after randomisation.
Surgical Debridement | Within the first 30 days after randomisation
  Total number of surgical debridements required by participants until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: sandramontedonico@gmail.com Montedonico, M.D., Study Director — Servicio de Cirugía Pediátrica, Hospital Carlos Van Buren, Valparaíso, Chile; Sebastián San Martín, Ph.D., Principal Investigator — Escuela de Medicina, Universidad de Valparaíso, Chile; Felipe Martínez, M.D., Principal Investigator — Escuela de Medicina, Universidad de Valparaíso, Chile
Locations (1):
- Hospital Carlos Van Buren, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selig HF, Lumenta DB, Giretzlehner M, Jeschke MG, Upton D, Kamolz LP. The properties of an "ideal" burn wound dressing--what do we need in daily clinical practice? Results of a worldwide online survey among burn care specialists. Burns. 2012 Nov;38(7):960-6. doi: 10.1016/j.burns.2012.04.007. Epub 2012 May 8. PMID 22571855
- [Background] Fairbairn NG, Randolph MA, Redmond RW. The clinical applications of human amnion in plastic surgery. J Plast Reconstr Aesthet Surg. 2014 May;67(5):662-75. doi: 10.1016/j.bjps.2014.01.031. Epub 2014 Jan 31. PMID 24560801
- [Background] Fraser JF, Cuttle L, Kempf M, Phillips GE, Hayes MT, Kimble RM. A randomised controlled trial of amniotic membrane in the treatment of a standardised burn injury in the merino lamb. Burns. 2009 Nov;35(7):998-1003. doi: 10.1016/j.burns.2009.01.003. Epub 2009 May 17. PMID 19447551
- [Background] Bilic G, Zeisberger SM, Mallik AS, Zimmermann R, Zisch AH. Comparative characterization of cultured human term amnion epithelial and mesenchymal stromal cells for application in cell therapy. Cell Transplant. 2008;17(8):955-68. doi: 10.3727/096368908786576507. PMID 19069637
- [Background] Vloemans AF, Hermans MH, van der Wal MB, Liebregts J, Middelkoop E. Optimal treatment of partial thickness burns in children: a systematic review. Burns. 2014 Mar;40(2):177-90. doi: 10.1016/j.burns.2013.09.016. Epub 2013 Nov 26. PMID 24290852
- See also: Chilean Ministry of Health Guidelines on the Management of the Burn Patient — http://www.enfermeriaaps.com/portal/guia-clinica-manejo-del-paciente-gran-quemado-minsal-chile-2016